CLINICAL TRIAL: NCT00181350
Title: Serial CT Scans for the Evaluation of Two Different Relocatable Fixation Systems in Fractionated Stereotactic Radiotherapy
Brief Title: Serial CT Scans in Fractionated Stereotactic Radiotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P03.1426L
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Brain Tumor
Keywords: brain tumor; fractionated stereotactic radiotherapy; fixationsystems; repositioning
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Relocatable fixation system

SUMMARY:
This study aims at providing a quantitative evaluation of the accuracy of two different fixation systems, where one system is also evaluated with two different set-ups.

DETAILED DESCRIPTION:
Stereotactic conformal radiotherapy (SCRT) combines the precision of the stereotactically guided tumor localisation and the radiobiological advantages of the fractionation. This implies an highly accurate repositioning of the isocenter of the cerebral target at the isocenter of the linac gantry and couch + 30 times. In the use of stereotactic conformal radiotherapy (SCRT) accuracy is the mainstay for the treatment of brain tumours. The reason are reduced safety margins around the tumour (or no margins) in order to reduce normal tissue dose.

This study aims at providing a quantitative evaluation of the accuracy of two different fixation systems, where one system is also evaluated with two different set-ups. The first approach will be based on the BrainLAB thermoplastic masque (the masque with (= standard fixation) and without a custom made bite-block), the second will use the BrianLAB relocatable frame with the bite- block and a home made fixation system.

Repositioning accuracy will be evaluated in a randomized manner patient-dependent and independent with the two fixation systems mentioned above.

The rationale is to determine the margins to define the planning target volume (PTV), it is necessary to know the set-up accuracy of the immobilization system. An overestimation of the PTV would lead to possible toxicity and an underestimation could lead to a geographical miss.

The main endpoint of this trial will be the accurate reproducibility of the fixation system evaluated by repeated CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of brain tumor
* Fractionated stereotactic radiotherapy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
CT scanning with a stereotactic lokalizer will take place once a week with a double scan (for 2 fixations) without contrast.

SECONDARY OUTCOMES:
No secondary measures.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitta Baumert, PHD, Principal Investigator — Maastricht Radiation Oncology
Locations (1):
- Maastricht Radiation Oncology, Heerlen, Limburg, Netherlands

REFERENCES:
- [Derived] Theelen A, Martens J, Bosmans G, Houben R, Jager JJ, Rutten I, Lambin P, Minken AW, Baumert BG. Relocatable fixation systems in intracranial stereotactic radiotherapy. Accuracy of serial CT scans and patient acceptance in a randomized design. Strahlenther Onkol. 2012 Jan;188(1):84-90. doi: 10.1007/s00066-011-0018-7. Epub 2011 Dec 24. PMID 22194025